CLINICAL TRIAL: NCT02511041
Title: Immunologic Effects of Supplemental Monosaccharide and Nucleoside Derivatives in Patients With Inherited Disorders of Glycosylation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150159; 15-I-0159
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-01-24

CONDITIONS: PGM3
Keywords: CDG; PGM3; Immune
MeSH Terms: interventions — Acetylglucosamine; Uridine

ARMS (1):
- 1 (Experimental): This is a prospective exploratory study of nucleoside and monosaccharide supplement-ation and its effect on immunologic parameters in patients with evidence of altered glycosylation and immunologic abnormalities. Up to 50 subjects will receive escalating doses of oralmonosaccharide until a maximum tolerated dose is found and maintained for 6 weeks. Then nucleosidesupplementation will be added and the maximum tolerated dose will continue for 12 weeks. Parameters of interest will be assessed at NIH every 8 weeks. Themaximum participation time for each subject is 252 days. We will begin with PGM3 deficient patients, who will self-administer oral GlcNAc followed by dual supplementation with GlcNAc and Uridine. The remaining subjects will then receive these supplements following the same step-wise approach.
  Interventions: Drug: N-Acetylglucosamine (GlcNAc); Drug: Uridine

INTERVENTIONS:
Drug: N-Acetylglucosamine (GlcNAc) — N-acetylglucosamine (GlcNAc), 2-acetamino-2-deoxy- <=-Dglucose, or 2- acetylamino)-2- deoxy-D-glucose, is a monosaccharide derivative of glucose. It is classified as dietary supplement in the United States. In general, it is a white and slightly sweet powder that melts at 221 degrees C. The solubility of GlcNAc is 25% in water, and 1% aqueous solutions are colorless and clear. GlcNAc is contraindicated for patients receiving warfarin, chemotherapy or diabetes drugs. As GlcNAc may interfere with blood sugar control during and after surgery, it is contraindicated during the two weeks prior to major surgery.
Drug: Uridine — Uridine 5 -monophosphate (UMP) disodium salt is a water soluble colorless crystalline powder which melts at 202oC.

SUMMARY:
Background:

- A congenital disorder of glycosylation (CDG) affects the cells that make up the organs and tissues. In these cells, sugar molecules do not properly attach to other molecules, which are the basic building blocks of cells. Changes in sugars seen in people with CDGs may lead to allergies and can change people s ability to fight infections. Researchers want to see if a sugar supplement called N-acetylglucosamine can help people with CDGs who have detectable changes in their immune systems.

Objective:

- To see if N-acetylglucosamine can help cells to function in a healthy way in people with CDGs.

Eligibility:

- People at least 2 years of age who have a CDG and immune system changes.

Design:

* Participants will be screened with a physical exam, medical history, and blood tests.
* One month later, participants will repeat the blood tests from the screening visit. Blood will be drawn on 2 different days in the same week.
* Participants will get N-acetylglucosamine supplements and instructions for how to take them. N-acetylglucosamine is a powder that can be added to food or drink.
* Participants will have a physical exam and blood tests every month during the study.
* After taking N-acetylglucosamine for about 4 months, participants will have more blood tests. They will get more N-acetylglucosamine supplements and a nucleoside supplement. The second supplement may be a powder or tablets that may be crushed and added to food. Participants will take both supplements for 5 months.
* After about 10 months in the study, participants will have 2 more visits in the same week for the same blood tests.

DETAILED DESCRIPTION:
Autosomal recessive hypomorphic loss-of-function mutations in phosphoglucomutase 3 (PGM3) have been shown to result in a novel congenital disorder of glycosylation (CDG) presenting with a hyper-IgE clinical phenotype. PGM3 is required for the biosynthesis of uridine diphosphate N-acetylglucosamine (UDP-GlcNAc), a critical building block for N- and O-linked glycans, which are essential for many immune pathways in humans. PGM3 deficient patients exhibit reduced UDP-GlcNAc levels, as well as both cell specific and global defects in N- and O-linked glycosylation, respectively. Understanding how glycosylation defects result in atopic diatheses and immune dysregulation will provide novel insight into their immunopathogenesis. Developing successful therapies in these patients may further provide novel targets or approaches to the treatment of allergic diseases in the general population.

Patients with other CDGs have shown dramatic clinical improvement when given oral supplementation with mannose and fucose. Among our patients with PGM3 deficiency, in vitro supplementation with the non-diabetogenic amino-sugar N-acetylglucosamine (GlcNAc) normalized intracellular UDP-GlcNAc and surface CTLA-4 expression. We therefore propose an exploratory study to provide up to 50 patients with exogenous GlcNAc and triacetyluridine with the objectives of assessing the effects on immune function and changes in cellular glycosylation patterns. We will begin with PGM3 patients who will self-administer sequential, escalating doses of oral GlcNAc and uridine ( UMP or TAU). Given our preliminary in vitro data, we hypothesize that supplementation will provide sufficient substrate to promote increased UDP-GlcNAc, restore N- and O-linked glycans, and improve immune function in PGM3 deficient patients.

Patients will self-administer oral GlcNAc 3 times per day beginning with 12.5 mg/kg/day and increasing the dose every 2 weeks. Once a maximum tolerated dose is found (less than or equal to 100 mg/kg/day), GlcNAc supplementation will continue for 6 weeks, at which point we will add oral uridine. We will titrate uridine to find its maximum tolerated dose

(less than or equal to 200 mg/kg/day) and continue dual dosing for an additional 12 weeks. If at the end this time period there has been no change in absolute lymphocyte count, supplementation will be stopped. The dietary supplements to be used in this study have very low toxicity and have been well-tolerated in studies of patients with colitis, galactosemia, Alzheimer s, multiple sclerosis, and in treatment of 5-fluorouracil overdose.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must have:

* Age greater than or equal to 2 years
* An inherited syndrome presenting with immunologic abnormalities and altered glycosylation detected using clinical tests evaluating N- and O-linked glycan by mass spectroscopy
* A local physician who is willing to follow the patient during the study period
* For females of childbearing potential, willingness to use a highly effective method of contraception (e.g., abstinence, intrauterine device [IUD]; oral contraceptives; diaphragms; or condom in combination with contraceptive foam, jelly, or cream; Norplant, contraceptive patch or cervical ring)
* Willingness to have samples stored for future research including genetic testing

EXCLUSION CRITERIA:

* Pregnant, breastfeeding, or intent to become pregnant
* Renal failure or chronic kidney disease requiring dialysis
* Uncontrolled asthma
* Abuse of drugs or alcohol as assessed during complete history and physical performed at the screening visit
* Current or recent participation in a clinical protocol which includes an intervention that, in the opinion of the investigator, may affect the results of the current study
* Use of medications that interact with N-acetylglucosamine including warfarin and medications for the treatment of cancer (antimitotic chemotherapy including etoposide, teniposide, and doxorubicin) and diabetes (including glimepiride, glyburide, insulin, pioglitazone, rosiglitazone, chlorpropamide, glipizide and tolbutamide).
* Planned major surgery during the study period requiring general anesthesia
* Any condition that in the opinion of the investigator places the patient at undue risk for being in the study
* Unwillingness or inability to comply with the need to have periodic blood tests to monitor possible side effects of supplementation, or other major requirements of this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06-30; Primary Completion 2017-01-24 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
In patients with evidence of altered glycosylation and immunologic abnormalities, to assess the effects of oral monosaccharides and nucleosides on: a) Absolute lymphocyte count | Monthly

SECONDARY OUTCOMES:
To assess the effects of oral monosaccharides and nucleosides on: e) Serum and secreted immunoglobulin levels f) Lymphocyte subsets, function, proliferation, and apoptosis g) Innate immune function h) Glycosylation patterns of serum and cellular... | Mid study Day 111 and end of study Day 252

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J Lyons, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Davis SD, Schaller J, Wedgwood RJ. Job's Syndrome. Recurrent, "cold", staphylococcal abscesses. Lancet. 1966 May 7;1(7445):1013-5. doi: 10.1016/s0140-6736(66)90119-x. No abstract available. PMID 4161105
- [Background] Buckley RH, Wray BB, Belmaker EZ. Extreme hyperimmunoglobulinemia E and undue susceptibility to infection. Pediatrics. 1972 Jan;49(1):59-70. No abstract available. PMID 5059313
- [Background] Holland SM, DeLeo FR, Elloumi HZ, Hsu AP, Uzel G, Brodsky N, Freeman AF, Demidowich A, Davis J, Turner ML, Anderson VL, Darnell DN, Welch PA, Kuhns DB, Frucht DM, Malech HL, Gallin JI, Kobayashi SD, Whitney AR, Voyich JM, Musser JM, Woellner C, Schaffer AA, Puck JM, Grimbacher B. STAT3 mutations in the hyper-IgE syndrome. N Engl J Med. 2007 Oct 18;357(16):1608-19. doi: 10.1056/NEJMoa073687. Epub 2007 Sep 19. PMID 17881745